CLINICAL TRIAL: NCT05386693
Title: Predicting Surgical Outcomes Following Neurectomy Based Upon Response to Local Anesthetic Injection in Chronic Groin Pain Patients
Brief Title: Surgical Outcomes Following Neurectomy Based Upon Response to Local Anesthetic Injection in Chronic Groin Pain
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, David Krpata, Principal Investigator, The Cleveland Clinic
Other Study IDs: 21-1176
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hernia, Inguinal; Chronic Postoperative Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ilioinguinal Nerve Block
  Interventions: Procedure: Ilioinguinal nerve block

INTERVENTIONS:
Procedure: Ilioinguinal nerve block — Local anesthetic injection of the ilioinguinal nerve. This is performed in the outpatient clinic.

SUMMARY:
The management of chronic pain after inguinal hernia surgery presents unique challenges. Ilioinguinal nerve blocks are often used in the initial treatment of this disease. This can often be followed by surgery, including neurectomy and/or hernia mesh removal. In an effort to identify preoperative predictors of postoperative outcomes following these surgical interventions the investigators devised a study to prospectively evaluate and correlate a patients pre-operative response to an ilioinguinal nerve block with their post-operative outcomes following surgery for chronic groin pain after inguinal hernia surgery.

DETAILED DESCRIPTION:
In the United States, 800,000 inguinal hernia repairs are performed annually, making it one of the most common surgical procedures.1,2 While major advancement has been gained in minimizing hernia recurrence, chronic pain after groin hernia repair remains the most common and significant complication of this surgery, drastically affecting patients' quality of life.3,4 Chronic pain has a substantial impact on physical, emotional, and cognitive function, on social and family life, and on the ability to work and secure an income 5. It has been reported that 5-10% of patients undergoing inguinal hernia repair develop postoperative chronic pain, the etiology of which remains unclear.6,7 Multiple behavioral, physical, and pharmacological interventions have shown positive results in treating chronic postoperative inguinal pain.8 Yet, some patients develop refractory pain severe enough to warrant removing the nerve tissue carrying the pain signal from the inguinal region, a procedure called neurectomy. While neurectomy provides an excellent outcome for some patients, others have no clear benefit from this surgery. 1,8-10 The challenge remains to identify which patients will gain the most advantage from neurectomy. Identifying patients who are least likely to benefit from the neurectomy will help spare them going through unnecessary pain and risk from the surgical intervention, reduce the cost of medical care, and focus efforts on other interventions that may provide better outcomes. This study aims to answer the question of whether or not pre-operative injection of an inguinal nerve predicts a patient's response to neurectomy.

Specific Aims

During the preoperative assessment for neurectomy, patients undergo a minor procedure involving injecting a local analgesic around the nerve, a nerve block. In this study, the investigators propose providing the patients with pain and quality of life questionnaires and tools to assess their baseline pain, response to the local analgesics, and response to the neurectomy procedure. The specific aims of the study are:

1. Evaluate the reliability of nerve block to predict patient response to neurectomy procedure:

   While nerve blocks have been frequently used as part of the preoperative assessment to neurectomy, the response from nerve block has not been correlated with post-neurectomy pain outcomes. The investigators intend to objectively assess pain relief in response to nerve block and neurectomy in this specific aim.

   The investigators hypothesized that patients who reported relief in response to nerve blocks would have pain relief from post neurectomy procedure, and patients who did not experience relief from nerve blocks will not have relief from post neurectomy procedure.
2. Evaluate the correlation between the extent of pain relief from nerve block to post neurectomy pain relief:

The Visual Assessment Scale (VAS) is a tool that provides a quantified assessment of pain. Assessing the pain with VAS before and after nerve block will provide a scale of change in pain level in response to the nerve block injection, the extent of which can be correlated with post neurectomy VAS to predict the outcome. The investigators hypothesize that patients with a greater improvement in pain level in response to nerve block have a higher chance of achieving pain relief with neurectomy than those with a low improvement in pain level from the nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of older)
* Chronic groin pain

Exclusion Criteria:

* Not a surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical intervention of chronic post-operative inguinal pain after inguinal hernia repair with or without mesh.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Change in pain levels | Baseline and 3 months after surgery
  Pain as measured with the Visual Analogue Scale (VAS) using a scale of 0 to 100; with 0 being the least amount of pain and 100 being the most amount of pain.
Change in pain levels | Baseline and 3 months after surgery
  Pain as measured with the Chronic Groin Pain Questionnaire which uses a Numeric Rating Scale (NRS). NRS uses a scale of 0 to 10; with 0 being the least amount of pain and 10 being the most amount of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No